CLINICAL TRIAL: NCT02349906
Title: Clinical Phase II Trial to Compare Treosulfan-based Conditioning Therapy With Busulfan-based Conditioning Prior to Allogeneic Haematopoietic Stem Cell Transplantation (HSCT) in Paediatric Patients With Non-malignant Diseases
Brief Title: Treosulfan-based Versus Busulfan-based Conditioning in Paediatric Patients With Non-malignant Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Collaborators: Celerion (Industry); Venn Life Sciences (Other); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC-FludT.16/NM
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Primary Immunodeficiencies; Inborn Errors of Metabolism; Haemoglobinopathies; Bone Marrow Failure Syndromes
Keywords: non-malignant diseases, allogeneic stem cell transplantation
MeSH Terms: conditions — Metabolism, Inborn Errors; Hemoglobinopathies; Bone Marrow Failure Disorders | interventions — treosulfan; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treosulfan (Experimental): One Treosulfan dose per day administered i.v. on three consecutive days (-6, -5 and -4); given over 2 hours as part of background conditioning prior to allogeneic stem cell transplantation.
  The dose has to be calculated as follows:
  If the BSA (m2) is equal or less than 0.3, the Treosulfan dose should be 10g/m2/day.
  If the BSA (m2) is greater than 0.3 and equal or less than 0.8, the Treosulfan dose should be 12g/m2/day.
  If the BSA (m2) is greater than 0.8, the Treosulfan dose should be 14g/m2/day.
  Interventions: Drug: Treosulfan
- Busulfan (Active Comparator): Total daily Busilvex dose (3.2 to 4.8 mg/kg/day, based on body weight) according to authorised dosage for children and adolescents administered i.v. as part of the background conditioning regimen on four consecutive days (days -7, -6, -5 and -4); given in 1, 2, or 4 portions per day according to the respective hospital's standard.
  Interventions: Drug: Busilvex

INTERVENTIONS:
Drug: Treosulfan
  Arms: Treosulfan
Drug: Busilvex
  Arms: Busulfan

SUMMARY:
The aim of the trial is to describe the safety and efficacy of intravenous (i.v.) Treosulfan compared to the conventional (myeloablative) dose of i.v. Busulfan, each administered as part of a standardised Fludarabine-containing conditioning regimen and to contribute to a PK model which permits - in conjunction with data comparing Treosulfan and Busulfan in adults with malignant diseases - to extend the use of Treosulfan in the paediatric population by extrapolating efficacy.

DETAILED DESCRIPTION:
The prospective clinical phase II protocol MC-FludT.16/NM is to be conducted to verify safety and efficacy of Treosulfan-based conditioning compared to Busulfan-based conditioning in paediatric patients. Based on the given clinical experience with either Treosulfan-based or Busulfan-based conditioning in combination with Fludarabine no increased risk for graft failure is expected in paediatric patients. A potential benefit for study patients is expected with respect to a probably low non-haematological toxicity of treatment compared to myeloablative TBI-based conditioning or high-dose Busulfan-based conditioning in combination with Cyclophosphamide.

However, the allogeneic HSCT procedure itself potentially involves serious risks with regard to severe or life-threatening conditions like graft versus host disease (GvHD) and/or infectious complications as well as graft failure.

In summary, the primary goal of this study is to evaluate the Treosulfan-based myeloablative conditioning regimen as an alternative in children and to contribute to the current PK model for Treosulfan to be able to finally give age (or body surface area [BSA]) dependent dose recommendations. The treatment regimens given in the protocol MC-FludT.16/NM are based on sufficient clinical safety and efficacy data. Considering the vital indication for allogeneic HSCT of the selected patient population, the risk-benefit assessment seems to be in favour of the study conduct.

Moreover, planned interim analyses will ensure the early identification of unexpected risks. Therefore, the conduct of the protocol MC-FludT.16/NM is considered reasonably justified.

ELIGIBILITY:
Inclusion Criteria:

1. Non-malignant disease indicated for first myeloablative allogeneic HSCT, including inborn errors of metabolism, primary immunodeficiencies, haemoglobinopathies and bone marrow failure syndromes.
2. First allogeneic HSCT.
3. Available matched sibling donor (MSD), matched family donor (MFD) or matched unrelated donor (MUD). For bone marrow (BM) and peripheral blood (PB) match is defined as at least 9/10 allele matches after four digit typing in human leucocyte antigen (HLA)-A, -B, -C, -DRB1 and DQB1 antigens. For umbilical cord blood (UCB) match is defined as at least 5/6 matches after two digit typing in HLA-A and -B and four digit typing in DRB1 antigens.

Exclusion Criteria:

1. Second or later HSCT.
2. HSCT from mismatched donor (less than 9/10 BM/peripheral blood stem cells (PBSC) or less than 5/6 matched cord donor).
3. Preterm newborn infants (<37 weeks gestational age) and term newborn infants aged 0 - 27 days at time of registration.
4. Obese paediatric patients with body mass index weight (kg)/[height (m)]² > 30 kg/m².
5. Diagnosis of Fanconi anaemia and other chromosomal breakage disorders, radiosensitivity disorders (deoxyribonucleic acid (DNA) Ligase 4, Cernunnos- X-ray repair cross-complementing protein 4 (XRCC4) like factor (XLF), Nijmegen Breakage Syndrome (NBS)) and Dyskeratosis Congenita.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2015-04; Primary Completion 2020-05-07 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Comparative evaluation of freedom from transplant (treatment)-related mortality (TRM), defined as death from any transplant-related cause from the day of first administration of study medication (day -7) until day +100 after HSCT. | day -7 to day +100

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Walter Sykora, MD and Prof, Principal Investigator — Hannover Medical University
Locations (21):
- University Hospital Motol, Dep. of Paediatric Haematology and Oncology, Prague, Czechia
- Germany (7):
  - Department of Pediatric Oncology & Hematology, Charite Berlin, Berlin
  - University Children's Hospital Essen Pediatric stem cell transplantation, Essen
  - University Hospital Frankfurt, Frankfurt am Main
  - Hannover Medical University, Dep. of Paediatrics, Paediatric Haematology and Oncology, Hanover
  - Heidelberg University Hospital, Heidelberg
  - University of Jena, Department of Pediatrics, Jena
  - Ulm, University Hospital, Clinic for Children and Adolescents, Ulm
- Italy (9):
  - SC Oncoematologia Pediatrica Ospedale Pediatrico Microcitemico "Antonio Cao" A.O. Brotzu, Cagliari
  - UOC Ematologia ed Oncologia Pediatrica con TMO AOU Policlinico Vittorio Emanuele, Catania
  - Reparto Trapianti Midollo Osseo Clinica Pediatrica Universitaria Fondazione MBBM-Ospedale San Gerardo, Monza
  - S.C. Oncoematologia Pediatrica Fondazione IRCCS Policlinico San Matteo, Pavia
  - Oncoematologia Pediatrica A.O. di Perugia Ospedale S. Maria della Misericordia, Perugia
  - U.O. Oncoematologia Pediatrica Azienda Ospedaliero Universitaria Pisana Ospedale S. Chiara, Pisa
  - Ospedale Bambino Gesu Roma, Rome
  - Ospedale Infantile Regina Margherita Torino, Turin
  - U.O.C. Oncoematologia Pediatrica Policlinico "G.B. Rossi" - AOUI Verona, Verona
- Poland (4):
  - Szpital Uniwersytecki im. dr Antoniego Jurasza, Bydgoszcz
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Dzieciecy Szpital Kliniczny im. A. Gebali w Lublinie, Lublin
  - Wroclaw Medical University, Department of Pediatric Hematology/Oncology and BMT, Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided